CLINICAL TRIAL: NCT05243407
Title: Sensing Physical Activity to Evaluate and Monitor a Routine Aftercare Program (SensE-M) - an Observational Study
Brief Title: Sensing Physical Activity to Evaluate and Monitor a Routine Aftercare Program (SensE-M)
Acronym: SensE-M
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Kliniken Valens (Unknown)
Responsible Party: Sponsor
Other Study IDs: V1
Record Dates: First submitted 2022-01-28; First posted 2022-02-17 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Disease With a Risk for Chronicity
Keywords: chronic disease; multiple sclerosis; cardiovascular disease; physical activity; activity tracker
MeSH Terms: conditions — Chronic Disease; Multiple Sclerosis; Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Conditions such as multiple sclerosis (MS) and cardiovascular diseases (CVDs) are severe and prevalent health conditions which decrease life expectancy and increase morbidity. Key symptoms of MS and CVDs include restrictions in physical activity which increase over time and severely affect individuals' quality of life. As such, promoting physical activity is at the core of state-of-the-art treatment for these diseases. However, any improvements in daily activity levels and physical fitness that may be achieved are typically challenging to maintain in daily life. Once back in their daily life environment, persons with chronic diseases face multiple barriers to physical activity such as fatigue, a less structured environment, or time restrictions associated with care responsibilities, employment, or the like.

Thus, a key challenge relates to the effective adaptation of physical activity-promoting routines and structures from the supportive rehab clinic environment to individuals' everyday lives. An example of an inpatient routine aftercare program which is designed to bridge this transition is the 'Stay with it'-program (Swiss German: 'Bliib dra'-program) developed by the Kliniken Valens. The program is designed to empower participants and promote self-efficacy and expertise - for example, in terms of self-management and self-monitoring skills. In addition, novel types of consumer-grade sensors, such as the Fitbit activity tracker, allow the assessment of a broad range of real-time activity- and sleep-related features and could complement the routine aftercare program. While these technical developments facilitate personalization and tailoring of health programs, it is often an untapped resource. However, health care professionals face time- and resource constraints. Consequently, any technical extensions of routine care programs tapping novel technical resources would need to be very scalable, streamlined, and efficient.

Objectives: The present project will thus explore the potential of leveraging novel technical development in the form of consumer-grade activity sensors to complement a routine aftercare program aiming to translate structures and skills from the inpatient stay to individuals' daily lives. Specifically, the project will examine whether and how concomitant evaluation of the 'Bliib dra'-program is effective, feasible, accepted, and sustainable. To this end, we will carefully examine the experiences and needs of both program participants and therapists and conclude with recommendations which can be generalized to similar types of routine aftercare programs which are conceptualized for adult persons for whom maintenance and increase of physical activity is vital (e.g., MS, CD, other chronic diseases and acute conditions that are at risk for a chronic course such as stroke).

DETAILED DESCRIPTION:
Primary hypothesis (hypothesis 1 - effective integration): The investigators hypothesize that integrating the Fitbit effectively into the program to measure activity goals will support program participants in pursuing their daily activity goals, particularly, once they have returned home. A prerequisite for the Fitbit's effective integration into individuals' daily lives will be the definition of activity goals which can be measured and tracked conveniently with the Fitbit.

Analysis plan: The analysis strategy will depend on the final sample size. Using a descriptive approach, the investigators will compute the difference between average daily activity after their return home and their predefined activity goals which have been defined as part of the 'Bliib dra'-program (e.g., active zone minutes of different intensity, steps per day) relative to previously agreed activity level goals. Furthermore, the investigators will examine participants' free text replies concerning challenges and facilitators in pursuing their activity goals in daily life and potential/difficulties of activity trackers in this regard. To extract relevant information, the investigators will evaluate Fitbit-related statements using natural language processing techniques.

Secondary hypothesis (hypothesis 2 - daily-life activity at home): Further, the investigators hypothesize that program participants will maintain a consistent and relatively stable level of physical activity.

Analysis plan: The analysis strategy will depend on the final sample size. The investigators will examine different activity level outcomes (e.g., active zone minutes, step count, high- /medium-intensity minutes) the time series data using descriptive and visual methods. If the sample size allows for more complex models, they will model physical activity over time and explore individual level-factors using a (multilevel) regression framework whereby controlling for individual-level factors. The investigators will investigate decline in activity levels defined as abrupt decrease or a steady decrease over an extended period of time (i.e., at least a week).

Exploratory: The investigators will further explore what challenges program participants and therapists experience, what they appreciate, and what they need to effectively integrate activity trackers such as the Fitbit device effectively into routine care program 'Bliib dra'. They will also explore how individual-level health measures (e.g., PROMIS-10) change over time.

Analysis plan: The investigators will examine therapists' and program participants' replies to the open questions using natural language processing techniques. With regard to the time series data, the analysis strategy will depend on the final sample size. They will examine the time series data using descriptive and visual methods. If the sample size allows for more complex models, the investigators will use a multivariable regression framework whereby controlling for individual-level factors.

ELIGIBILITY:
Inclusion criteria are:

* Female and male inpatients who are for an inpatient stay at Kliniken Valens and participate in the 'Bliib dra'-program while the study is ongoing. The 'Bliib dra'-program is conceptualized for adult persons who have a diagnosis of MS, a cardiovascular disease, diabetes, stroke, or hypertension.
* Provision of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are at Kliniken Valens for an inpatient rehabilitation stay and participate in the 'Bliib dra'-program are eligible for the study. Program participants that are interested in the study will be provided with the study information sheet, detailing study aims and procedure. We will enroll patients if they agree to participate and provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Active zone minutes (Fitbit) | through study completion, on average 4 months
  Rate of energy expended during an activity : rate of energy expended during rest
Step count (Fitbit) | through study completion, on average 4 months
Minutes spent in activity intensity levels (high, moderate, low; Fitbit) | through study completion, on average 4 months
Heart rate (Fitbit) | through study completion, on average 4 months
Answers to open questions for program participants and therapists regarding the implementation of the 'Stay with it'-program as well as their experience with the Fitbit | prior to program start, at clinic discharge (i.e., on average after 1 month), and 3-month follow-up

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System - Global 10 (PROMIS-10) | at clinic admission, at clinic discharge (i.e., on average after 1 month), and 3-month follow-up
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | prior to program start, at clinic discharge (i.e., on average after 1 month), and 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Viktor von Wyl, Prof. Dr., Principal Investigator — Institute for Implementation Science in Health Care, University of Zurich
Locations (1):
- Kliniken Valens, Valens, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams V, Linke A. Impact of exercise training on cardiovascular disease and risk. Biochim Biophys Acta Mol Basis Dis. 2019 Apr 1;1865(4):728-734. doi: 10.1016/j.bbadis.2018.08.019. Epub 2018 Aug 28. PMID 30837069
- [Background] Brouns B, van Bodegom-Vos L, de Kloet AJ, Tamminga SJ, Volker G, Berger MAM, Fiocco M, Goossens PH, Vliet Vlieland TPM, Meesters JJL. Effect of a comprehensive eRehabilitation intervention alongside conventional stroke rehabilitation on disability and health-related quality of life: A pre-post comparison. J Rehabil Med. 2021 Mar 5;53(3):jrm00161. doi: 10.2340/16501977-2785. PMID 33369683
- [Background] Kalb R, Brown TR, Coote S, Costello K, Dalgas U, Garmon E, Giesser B, Halper J, Karpatkin H, Keller J, Ng AV, Pilutti LA, Rohrig A, Van Asch P, Zackowski K, Motl RW. Exercise and lifestyle physical activity recommendations for people with multiple sclerosis throughout the disease course. Mult Scler. 2020 Oct;26(12):1459-1469. doi: 10.1177/1352458520915629. Epub 2020 Apr 23. PMID 32323606
- [Background] Katzan I, Schuster A, Kinzy T. Physical Activity Monitoring Using a Fitbit Device in Ischemic Stroke Patients: Prospective Cohort Feasibility Study. JMIR Mhealth Uhealth. 2021 Jan 19;9(1):e14494. doi: 10.2196/14494. PMID 33464213
- [Background] Murray E, Treweek S, Pope C, MacFarlane A, Ballini L, Dowrick C, Finch T, Kennedy A, Mair F, O'Donnell C, Ong BN, Rapley T, Rogers A, May C. Normalisation process theory: a framework for developing, evaluating and implementing complex interventions. BMC Med. 2010 Oct 20;8:63. doi: 10.1186/1741-7015-8-63. PMID 20961442
- [Background] Silveira SL, Motl RW. Activity monitor use among persons with multiple sclerosis: Report on rate, pattern, and association with physical activity levels. Mult Scler J Exp Transl Clin. 2019 Nov 9;5(4):2055217319887986. doi: 10.1177/2055217319887986. eCollection 2019 Oct-Dec. PMID 31741742
- [Background] Van Geel F, Geurts E, Abasiyanik Z, Coninx K, Feys P. Feasibility study of a 10-week community-based program using the WalkWithMe application on physical activity, walking, fatigue and cognition in persons with Multiple Sclerosis. Mult Scler Relat Disord. 2020 Jul;42:102067. doi: 10.1016/j.msard.2020.102067. Epub 2020 Apr 18. PMID 32371377